CLINICAL TRIAL: NCT03527524
Title: Effects of Core Stabilization Exercises With and Without Ball on Pain, Functional Disability and Level of Lumbar Stability in Patients With Non-specific Chronic Low Back Pain
Brief Title: Effect of Exercises on Pain, Functional Disability and Lumbar Stability in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MahidolU_Wunpen1
Record Dates: First submitted 2017-01-05; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Exercise
Keywords: exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise with ball (Experimental): The participant in core stabilization exercise with ball group performed 12 training sessions of the core stabilization exercises, 3 days/week for 4 weeks. Each exercise took 15 times/set and each participant did it repeatedly for 3 sets and rested 1 minute between sets. The total time of core stabilization exercise was 20 minutes and assessment time was 10 minutes.
  Interventions: Other: exercise with ball
- exercise without ball (Other): The participant in core stabilization exercise without ball group performed 12 training sessions of the core stabilization exercises, 3 days/week for 4 weeks. Each exercise took 15 times/set and each participant did it repeatedly for 3 sets and rested 1 minute between sets. The total time of core stabilization exercise was 20 minutes and assessment time was 10 minutes.
  Interventions: Other: exercise without ball

INTERVENTIONS:
Other: exercise with ball — exercise with ball
  Arms: exercise with ball
Other: exercise without ball — exercise without ball
  Arms: exercise without ball

SUMMARY:
The purposes of this study are to compare the effects of core stabilization exercises on pain intensity, functional disability and lumbar stability between using and not using the Swiss ball in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
For Patient Registries:

The participant was screened for inclusion criteria and was asked to sign the informed consent prior to participate. A randomized control trial was performed with participants randomly divided into one of the two treatment groups: core stabilization exercise with ball and core stabilization exercise without ball by using sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female with low back pain (LBP) > 3 months
2. Body mass index (BMI) = 18-25 kg/m2
3. Non-specific LBP (pain at the lower lumbar between costal margin but not below gluteal fold)
4. Willing and able to perform exercise programs
5. No cognitive impairment
6. Age at least 19 years

Exclusion Criteria:

1. Having experiences in the core stabilization exercise and Swiss ball exercises
2. Past history of back and abdomen surgery
3. Recent fractures of spine, hip or lower limb
4. Current use of steroids or any other drugs for resolving back pain
5. Red flags (fractures, cancer, infection, cauda equine syndrome)
6. Pregnancy
7. Neuromuscular or respiratory disorders
8. Rheumatologic disorders
9. Hip and knee stiffness
10. Pain intensity > 60 of 100 mm assessed by the VAS

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain scale | 4 weeks
  a 0-100 mm of horizontal line (Visual analog scale) assessing pain intensity - reported the distance measured in millimeters from the left hand side of this line to the point that participant marked

SECONDARY OUTCOMES:
Questionnaire scores of functional disability measure | 4 weeks
  Thai modified Oswestry Disability Low Back Pain Disability Questionnaire
Levels of lumbar stability | 4 weeks
  isometric abdominal contraction assessing lumbar stability

CONTACTS AND LOCATIONS:
Overall Officials: Apinkarn Jaroenlarp, MSc, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No